CLINICAL TRIAL: NCT00125190
Title: Recombinant Human Insulin-Like Growth Factor (rhIGF-1) Treatment of Short Stature Associated With Primary IGF-1 Deficiency: A Multi-Center, Open Label, Concentration-Controlled Study
Brief Title: Recombinant Human Insulin-Like Growth Factor (rhIGF-1) Treatment of Short Stature Associated With IGF-1 Deficiency
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS308; 2019-001095-11 (EudraCT Number)
Record Dates: First submitted 2005-07-27; First posted 2005-07-29 (Estimated); Results first posted 2010-04-15 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Insulin-Like Growth Factor-1 Deficiency; Growth Disorders
Keywords: Primary IGF-1 Deficiency; IGF-1
MeSH Terms: conditions — Growth Disorders | interventions — mecasermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rhIGF-1 QD (Experimental): Subjects received subcutaneous injection (SC) injections of rhIGF-1 once a day.
  Interventions: Drug: rhIGF-1 (mecasermin) for a period of 86 weeks

INTERVENTIONS:
Drug: rhIGF-1 (mecasermin) for a period of 86 weeks — Once a day rhIGF-1 injections

SUMMARY:
This study is intended to assess the effects of once daily dosing of recombinant human insulin-like growth factor (rhIGF-1) in increasing height velocity.

DETAILED DESCRIPTION:
Growth failure associated with primary IGF-1 deficiency (IGFD). Primary IGFD is a term that has been used to describe patients with intrinsic cellular defects in growth hormone (GH) action. In this protocol, primary IGFD is defined as short stature (<-2 standard deviations [SDs] below the mean for age and gender), and abnormal serum IGF-1 (<-2 SDs below the mean for age and gender).

The trial is an open-label, concentration-controlled trial conducted at up to 20 centers throughout the United States.

ELIGIBILITY:
Inclusion Criteria:

* Chronological age ≥ 3
* Chronological age or bone age ≤ 12 for boys and ≤ 11 for girls
* Prepubertal at Visit 1
* Height SD score of < -2
* IGF-1 SD score of < -2

Exclusion Criteria:

* Prior treatment with GH, IGF-1, or other growth-influencing medications
* Growth failure associated with other identifiable causes (e.g., syndromes, chromosomal abnormality)
* Chronic illness such as diabetes, cystic fibrosis, etc.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Study Director, M.D., Study Director — Ipsen
Locations (1):
- Ipsen, Brisbane, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a open-label, multi-center and single-arm study conducted at 12 investigational sites (11 active) between 12 January 2005 and 14 January 2009. A total of 45 subjects were enrolled in this study.
Pre-assignment Details: The screening period consisted of two-staged clinic visits for up to 6 weeks, followed by an open-label treatment period of 86 weeks.
Groups:
- rhIGF-1 QD: During the treatment phase (Day 1 to Week 86), subjects received subcutaneous (SC) injections of rhIGF-1 at an initial dose of 60 microgram per kilogram (mcg/kg) once daily (QD) starting on Day 1 (Visit 3). From Week 2 (Visit 4) subsequent dose adjustments were made in order to achieve the target serum IGF-1 concentration for the subject's age and sex. The maximum dose in any circumstance was 240 mcg/kg/day.
Period: Overall Study
Arm/Group | rhIGF-1 QD
Started | 45
Completed 34 Weeks of Study | 43
Completed | 30
Not Completed | 15
Not completed — Subject/Parent Decision | 7
Not completed — Non-compliance | 2
Not completed — Adverse Event | 1
Not completed — Other | 1
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) population included all treated subjects.
Groups:
- rhIGF-1 QD: During the treatment phase (Day 1 to Week 86), subjects received SC injections of rhIGF-1 at an initial dose of 60 mcg/kg QD starting on Day 1 (Visit 3). From Week 2 (Visit 4) subsequent dose adjustments were made in order to achieve the target serum IGF-1 concentration for the subject's age and sex. The maximum dose in any circumstance was 240 mcg/kg/day.
Arm/Group | rhIGF-1 QD
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.7 (2.8)
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 36
  Adolescents (12-17 years) | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 38
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 1
  Hispanic | 12
  White | 31
  Other | 1
Body Mass Index Standard Deviation (SD) Score [Mean (Standard Deviation); unit: SDs] | -0.4 (0.7)
Bone Age Imputed [Mean (Standard Deviation); unit: years] | 7.2 (2.6)
Height for Age SD Score [Mean (Standard Deviation); unit: SDs] | -2.7 (0.6)
IGFBP-3 SD Score [Mean (Standard Deviation); unit: SDs] | -0.7 (1.0)
IGF-1 SD Score [Mean (Standard Deviation); unit: SDs] | -2.6 (0.5)
Maximum Stimulated GH [Mean (Standard Deviation); unit: nanogram per milliliter] | 20.5 (9.9)
Weight for Age SD Score [Mean (Standard Deviation); unit: SDs] | -2.3 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Height Velocity From Pretreatment (Week 0) to Week 34
Description: Height was measured standing without shoes as the average of three measurements by the same observer using identical technique with a Harpenden or other wall mounted stadiometer. The subject was repositioned between each measurement. Height velocity during an interval of time is defined as the change in height during the time interval divided by the duration of the time interval. Missing Week 34 heights were imputed using the last height SD score carried forward.
Time Frame: Pretreatment to Week 34
Population: The ITT population included all treated subjects.
Measure: Mean (Standard Deviation); unit: centimeters per year (cm/yr)
Arm/Group | rhIGF-1 QD
Number analyzed (Participants) | 45
centimeters per year (cm/yr) | 7.0 (1.5)

2. Primary Outcome: Height Velocity From Week 34 to 86
Description: Height was measured standing without shoes as the average of three measurements by the same observer using identical technique with a Harpenden or other wall mounted stadiometer. The subject was repositioned between each measurement. Height velocity during an interval of time is defined as the change in height during the time interval divided by the duration of the time interval. Missing Week 86 heights were imputed using the last height SD score carried forward.
Time Frame: Week 34 to 86
Population: The ITT population included all treated subjects. Only subjects in the ITT population who continued past Week 34 were included in the analysis.
Measure: Mean (Standard Deviation); unit: cm/yr
Arm/Group | rhIGF-1 QD
Number analyzed (Participants) | 40
cm/yr | 6.7 (1.8)

3. Secondary Outcome: Change in Height SD Score From Pretreatment to Week 34
Description: Height was measured standing without shoes as the average of three measurements by the same observer using identical technique with a Harpenden or other wall mounted stadiometer. The subject was repositioned between each measurement. The SD score is calculated as the subject value minus the mean divided by the standard deviation. The mean and the standard deviation vary depending on the age and sex of the child.
Time Frame: Pretreatment and Week 34
Population: The ITT population included all treated subjects.
Measure: Mean (Standard Deviation); unit: SDs
Arm/Group | rhIGF-1 QD
Number analyzed (Participants) | 45
SDs | 0.21 (0.20)

4. Secondary Outcome: Change in Height SD Score From Pretreatment to Week 86
Description: Height was measured standing without shoes as the average of three measurements by the same observer using identical technique with a Harpenden or other wall mounted stadiometer. Subjects were repositioned between each measurement. The SD score is calculated as the patient value minus the mean divided by the standard deviation. The mean and the standard deviation vary depending on the age and sex of the child.
Time Frame: Pretreatment and Week 86
Population: The ITT population included all treated subjects. Only subjects who had both pretreatment and Week 86 measurements were included in the analysis.
Measure: Mean (Standard Deviation); unit: SDs
Arm/Group | rhIGF-1 QD
Number analyzed (Participants) | 40
SDs | 0.45 (0.39)

5. Secondary Outcome: Change in Bone Age From Pretreatment to Week 86 Minus Change in Chronological Age
Description: Plain X-rays of the left hand and wrist were exposed for bone age appraisal. The films were sent to a central facility for standardized evaluation.
Time Frame: Pretreatment to Week 86
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: years
Arm/Group | rhIGF-1 QD
Number analyzed (Participants) | 30
years | 0.2 (0.68)

6. Secondary Outcome: Percent Change in Serum Concentration of IGFBP-1, IGFBP-2 and IGFBP-3 From Pretreatment to Week 86
Description: Growth factor panels for measuring IGFBP-1, IGFBP-2 and IGFBP-3 were evaluated from screening and at each study visit up to Week 86. Inter-quartile range (Q1-Q3) is 10th to 90th percentile.
Time Frame: Pretreatment and Week 86
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | rhIGF-1 QD
Number analyzed (Participants) | 29
percent change
  IGFBP-1 | -89.6 [-96 to -13]
  IGFBP-2 | 37.9 [-25 to 227]
  IGFBP-3 | 0 [-27 to 48]

7. Secondary Outcome: Percent Change in Serum Concentration of ALS From Pretreatment to Week 86
Description: Growth factor panels for measuring ALS were evaluated from screening and at each study visit up to Week 86. Inter-quartile range (Q1-Q3) is 10th to 90th percentile.
Time Frame: Pretreatment and Week 86
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | rhIGF-1 QD
Number analyzed (Participants) | 29
percent change | -7.7 [-36 to 42]

8. Post Hoc Outcome: Increase in Height Velocity From Pretreatment to Week 34
Description: as for outcome 1
Time Frame: Pretreatment to Week 34
Population: Completer population included all subjects who remained on study to Week 86. Subjects who completed Week 34 were included in the analysis.
Measure: Mean (Standard Deviation); unit: cm/yr
Arm/Group | rhIGF-1 QD
Number analyzed (Participants) | 43
cm/yr | 1.3 (3.56)

9. Post Hoc Outcome: Increase in Height Velocity From Pretreatment to Week 86
Description: as for outcome 2
Time Frame: Pretreatment to Week 86
Population: Completer population included all subjects who remained on study to Week 86.
Measure: Mean (Standard Deviation); unit: cm/yr
Groups:
- rhIGF-1 QD: During the treatment phase, subjects received subcutaneous (SC) injections of rhIGF-1 at an initial dose of 60 µg/kg QD, with subsequent dose adjustments made in order to achieve the target serum IGF-1 concentration for the subject's age and sex. The maximum dose in any circumstance was 240 mcg/kg/day.
Arm/Group | rhIGF-1 QD
Number analyzed (Participants) | 30
cm/yr | 1.3 (3.58)

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected from Day 1 to Week 86 (approximately 21 months).
Arm/Group | rhIGF-1 QD
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 2/45
Other Adverse Events (participants affected / at risk) | 41/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhIGF-1 QD (N=45)
Gastroenteritis (Infections and infestations) | 1 (1)
Arnold-Chiari Malformation (Congenital, familial and genetic disorders) | 1 (1)
Syringomyelia (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhIGF-1 QD (N=45)
Abdominal Pain (Gastrointestinal disorders) | 3 (3)
Abdominal Pain Upper (Gastrointestinal disorders) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 5 (6)
Stomach Discomfort (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 18 (21)
Injection Site Bruising (General disorders) | 3 (5)
Pyrexia (General disorders) | 14 (18)
Gastroenteritis (Infections and infestations) | 6 (8)
Gastroenteritis Viral (Infections and infestations) | 3 (4)
Influenza (Infections and infestations) | 5 (6)
Nasopharyngitis (Infections and infestations) | 3 (5)
Otitis Media (Infections and infestations) | 5 (7)
Sinusitis (Infections and infestations) | 4 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 13 (24)
Viral Infection (Infections and infestations) | 7 (13)
Hypoglycaemia (Metabolism and nutrition disorders) | 5 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8)
Headache (Nervous system disorders) | 18 (32)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (13)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other